CLINICAL TRIAL: NCT03835793
Title: Favourable and Unfavourable Health Effects of Risk-Reducing Salpingo-Oophorectomy in Women With a High Genetic Risk of Ovarian Cancer
Brief Title: Health After eaRly Menopause Due to Oophorectomy
Acronym: HARMOny
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Cancer Society (Other); Erasmus Medical Center (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: M18HAR
Record Dates: First submitted 2018-09-19; First posted 2019-02-11 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Surgical Menopause; BRCA1 Mutation; BRCA2 Mutation; Cardiovascular Diseases; Bone Mineral Density; Cognitive Decline; Quality of Life; Menopause Surgical
Keywords: long-term; premature ovarian insufficiency
MeSH Terms: conditions — Cardiovascular Diseases; Cognitive Dysfunction; Primary Ovarian Insufficiency | interventions — Blood Specimen Collection; Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Optional for studyparticipants is to collect and store DNA in a blood Biobank.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early-RRSO: * RRSO before the age of 45 years
  * RRSO was done 10 or more years ago
  Interventions: Diagnostic Test: CAC-score
- Late-/non-RRSO group: * Natural menopause ≥ 50 years of age
  * No RRSO ≤ age of 55
  * No treatment-induced menopause ≤ 50 years of age
  Interventions: Diagnostic Test: CAC-score

INTERVENTIONS:
Diagnostic Test: CAC-score — Testing for possible unfavourable health effects of early surgical menopause
  Other Names: Blood sampling; DXA-scan; Vertebral Fracture Assessment; Online cognition test (Amsterdam Cognition Scale); Quality of life questionnaire

SUMMARY:
Risk-Reducing Salpingo-Oophorectomy (RRSO) at the age of 35 to 45 years is recommended for women with a high genetic risk for ovarian cancer. While this procedure decreases the risk of ovarian cancer by 80-96%, it also results in an immediate menopause. Current research on potential adverse effects of premenopausal risk-reducing salpingo-oophorectomy, such as increased risk of cardiovascular disease, compromised bone health, cognitive dysfunction and reduced quality of life, is limited, mostly due to short follow up.

The investigators will conduct a multicenter cross-sectional study nested in a cohort of BRCA mutation carriers from 8 Dutch centers for hereditary cancer. Eligible participants are women who underwent RRSO before the age of 45. The participants will be frequency-matched on current age with women above the age of 55 without RRSO or with RRSO after the age of 55. Participants will complete an online questionnaire containing various questions about lifestyle, medical history, risk factors for cardiovascular disease, bone health, cognition and quality of life. Participants will be asked to visit one of the participating hospitals for a blood test, a cardiovascular assessment and a DEXA scan for determining bone mineral density. Afterwards participants will be requested to perform the online Amsterdam Cognition Scale.

DETAILED DESCRIPTION:
Rationale: Women at high genetic risk of ovarian cancer are advised to undergo risk-reducing salpingo-oophorectomy (RRSO) at ages 35-45 years. Currently, in the Netherlands ~500 women/ year opt for RRSO, which minimizes ovarian cancer risk and may decrease breast cancer (BC) risk as well, due to reduced gonadal hormone levels. Besides favorable effects of RRSO on ovarian cancer and, potentially, BC risk, RRSO induces immediate menopause, which may have unfavorable long-term health consequences. Early menopause has been associated with increased risks of cardiovascular disease (CVD), lower bone mineral density (BMD), cognitive impairment, and decreased quality of life. Current evidence regarding these health effects is mainly based on women with a natural early menopause, and it is unknown whether these results hold for women undergoing RRSO at early premenopausal ages.

Objective: The investigators will investigate long-term health effects of premenopausal RRSO on (subclinical) cardiovascular status, BMD, cognition and quality of life.

Study design: the investigators will assess long-term health effects of RRSO in a cross-sectional study, among 500 women who underwent premenopausal RRSO compared to 250 women of the same age without RRSO (or with RRSO after age 55). Eligible women will be invited to participate in a screening program assessing cardiovascular status, bone mineral density, cognitive functioning and quality of life.

Study population: Women are eligible for the premenopausal RRSO group if:

* RRSO before the age of 45 years;
* RRSO was done 10 or more years ago; Women are eligible for the comparison group without premenopausal RRSO if the participant did not undergo RRSO before the age of 55 years, and did not have a natural or therapy induced menopause before age 50.

Primary study outcome: To study long-term effects of premenopausal RRSO on:

* (subclinical) CVD
* BMD
* Cognition

Secondary study outcome: To study long-term effects of premenopausal RRSO on:

* Quality of life
* Urogenital problems
* Cardiovascular risk factors

Furthermore, the investigators will examine the influence of age at RRSO, time since RRSO, hormone replacement therapy (HRT), carrier ship of a BRCA1 or BRCA2 mutation and BC history on the outcome.

The obtained knowledge will assist physicians in counselling women with high ovarian cancer risk and help them to make well-informed decisions.

ELIGIBILITY:
Inclusion Criteria:

* RRSO before age 45
* RRSO after age 55
* no RRSO

Exclusion Criteria:

* metastatic disease
* Premature ovarian insufficiency
* Physical or mental problems interfering with a outpatient visit
* nonbioabsorbable cardiac stent
* insufficient understanding of the Dutch language

Min Age: 55 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — In order to be eligible the ovaries have been removed.
Study Population: Women are eligible if they underwent RRSO before age 45 and the RRSO was done 10 or more years ago (early RRSO group) and women are eligible as control group if they did not undergo RRSO, or underwent RRSO after age 55 while reaching natural menopause after the age of 50 years. The comparison group will be frequency-matched with the RRSO group on categories of calendar year of birth, and breast cancer history. For each patient with breast cancer, the investigators will perform individual matching accounting for age at breast cancer diagnosis and carrier status. For the early RRSO group the investigators select women who underwent RRSO at least 10 years ago and are currently older than 55 years because the investigators expect subclinical atherosclerosis not to manifest earlier.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
What is the prevalence of atherosclerotic diseases in women with RRSO compared to women with a high genetic risk of ovarian cancer with a natural menopause as assessed by coronary artery calcium scoring in agatston units | 4 years
  Due to the lack of estrogen we expect more atherosclerotic diseases.
What is the prevalence of atherosclerotic diseases in women with RRSO compared to women with a high genetic risk of ovarian cancer with a natural menopause as assessed by pulse wave velocity in meters/second | 4 years
  Due to the lack of estrogen we expect more atherosclerotic diseases.
What is the prevalence of atherosclerotic diseases in women with RRSO compared to women with a high genetic risk of ovarian cancer with a natural menopause as assessed by high-sensitive CRP in miligram/liter | 4 years
  Due to the lack of estrogen we expect more atherosclerotic diseases.
What is the prevalence of atherosclerotic diseases in women with RRSO compared to women with a high genetic risk of ovarian cancer with a natural menopause as assessed by high-sensitive cardial Troponine T in microgram/liter | 4 years
  Due to the lack of estrogen we expect more atherosclerotic diseases.
What is the prevalence of osteoporosis in women with a premenopausal RRSO compared to women with a high genetic risk of ovarian cancer with a natural menopause as assessed by dual-energy X-ray absoptiometry in T- and Z-scores | 4 years
  Loss of estrogen can result in more activity of osteoclasts and less activity of osteoblasts, The DXA-scan is corrected for age, with lower values representing a worse outcome
What is the prevalence of osteoporosis in women with a premenopausal RRSO compared to women with a high genetic risk of ovarian cancer with a natural menopause as assessed by instant vertebral assessment | 4 years
  Loss of estrogen can result in more activity of osteoclasts and less activity of osteoblasts
What is the prevalence of osteoporosis in women with a premenopausal RRSO compared to women with a high genenetic risk of ovarian cancer with a natural menopause as assessed by beta-CTX in picogram/mililiter | 4 years
  Loss of estrogen can result in more activity of osteoclasts and less activity of osteoblasts
What is the prevalence of osteoporosis in women with a premenopausal RRSO compared to women with a high genenetic risk of ovarian cancer with a natural menopause as assessed by P1NP in miligram/liter | 4 years
  Loss of estrogen can result in more activity of osteoclasts and less activity of osteoblasts
What is the prevalence of cognitive decline in women with RRSO compared to women with a natural menopause as assessed by the Amsterdam Cognition Scan | 4 years
  There are some studies suggesting that an early menopause has an influence on cognition

SECONDARY OUTCOMES:
Quality of life after a premenopausal RRSO compared to women from families with a high genetic risk of ovarian cancer with a natural menopause as assessed by validated questionnaires such as the SF-36 | 4 years
  How do women with a premenopausal RRSO experience their life. The SF-36 questionnaire ranges from 36 to 149, with higher values representing a worse outcome
Quality of life after a premenopausal RRSO compared to women from families with a high genetic risk of ovarian cancer with a natural menopause as assessed by validated questionnaires such as the EORTC-QLQ BR23. | 4 years
  How do women with a premenopausal RRSO experience their life. We measure the body image using the EORTC QLQ BR23, with ranges from 2 to 8, with higher values representing a worse outcome
Quality of life after a premenopausal RRSO compared to women from families with a high genetic risk of ovarian cancer with a natural menopause as assessed by validated questionnaires such as the FACT-ES | 4 years
  How do women with a premenopausal RRSO experience their life. The FACT-ES questionnaire ranges from 0 to 76, with higher values representing a worse outcome
What is the prevalence of urogenital problems in women with a RRSO compared to women with a natural menopause as assessed by validated questionnaires such as the SAQ | 4 years
  Have women with a premenopausal RRSO more urogenital complaints due to longer duration of estrogen deficiency.
  The SAQ questionnaire scale has questions with different weights as described in Thirlaway et al. 1996
What is the prevalence of urogenital problems in women with a RRSO compared to women with a natural menopause as assessed by validated questionnaires such as the UDI-6 | 4 years
  Have women with a premenopausal RRSO more urogenital complaints due to longer duration of estrogen deficiency.
  The UDI-6 questionnaire scale has a range from 0 to 18, with higher values representing a worse outcome
What is the prevalence of urogenital problems in women with a RRSO compared to women with a natural menopause as assessed by validated questionnaires such as the IIQ-7 | 4 years
  Have women with a premenopausal RRSO more urogenital complaints due to longer duration of estrogen deficiency.
  The IIQ-7 questionnaire scale has a range from 0 to 24, with higher values representing a worse outcome
What is the prevalence of cardiovascular risk factors in women with RRSO compared to women with a high genetic risk of ovarian cancer as assessed by a questionnaire. | 4 years
  Are some risk factors for cardiovascular disease more prevalent in women with a premenopausal RRSO

OTHER OUTCOMES:
What is the effect of premenopausal RRSO on risk of (contralateral) breast cancer and breast cancer-specific survival as assessed in a prospective setting within a well established cohort. | 4 years
  we will study the effect of RRSO on BC, contralateral breast cancer and ovarian cancer risk and prognosis after BC/ovarian cancer

CONTACTS AND LOCATIONS:
Overall Officials: Flora E van Leeuwen, Phd, Principal Investigator — NKI-AvL
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beekman MJ, Terra L, Stuursma A, Heemskerk-Gerritsen BAM, van Lennep JER, van Beurden M, van Doorn LC, de Hullu JA, van Dorst EBL, Mom CH, Slangen BFM, Mitea C, Slart RHJA, Snoeren MM, Stokkel MP, Verberne HJ, de Keizer B, Korse CM, Gaarenstroom KN, van Engelen K, van der Kolk LE, Collee JM, Wevers MR, Ausems MGEM, Berger LPV, Garcia EBG, van Asperen CJ, Hooning MJ, Maas AHEM, Mourits MJE, van Leeuwen FE, Zillikens MC. Long-term effects of premenopausal risk-reducing salpingo-oophorectomy on bone mineral density. Osteoporos Int. 2025 Nov;36(11):2307-2317. doi: 10.1007/s00198-025-07679-8. Epub 2025 Oct 4. PMID 41045325
- [Derived] Beekman MJ, Terra L, Roeters van Lennep JE, Heemskerk-Gerritsen BAM, van Beurden M, van Doorn HC, de Hullu JA, van Dorst EBL, Mom CH, Slangen BFM, Mourits MJE, Gaarenstroom KN, van Engelen K, van der Kolk LE, Collee JM, Wevers MR, Ausems MGEM, Berger LPV, Gomez Garcia EB, van Asperen CJ, Hooning MJ, van Leeuwen FE, Maas AHEM. No increased arterial stiffness after premenopausal risk-reducing salpingo-oophorectomy (RRSO). Maturitas. 2025 Jun;197:108265. doi: 10.1016/j.maturitas.2025.108265. Epub 2025 Apr 11. PMID 40262388
- [Derived] Terra L, Beekman MJ, Engelhardt EG, Heemskerk-Gerritsen BAM, van Beurden M, Roeters van Lennep JE, van Doorn HC, de Hullu JA, Van Dorst EBL, Mom CH, Slangen BFM, Gaarenstroom KN, van der Kolk LE, Collee JM, Wevers MR, Ausems MGEM, Van Engelen K, van de Beek I, Berger LPV, van Asperen CJ, Gomez Garcia EB, Maas AHEM, Hooning MJ, Aaronson NK, Mourits MJE, van Leeuwen FE. Sexual functioning more than 15 years after premenopausal risk-reducing salpingo-oophorectomy. Am J Obstet Gynecol. 2023 Apr;228(4):440.e1-440.e20. doi: 10.1016/j.ajog.2022.11.1289. Epub 2022 Nov 17. PMID 36403862
- [Derived] Terra L, Hooning MJ, Heemskerk-Gerritsen BAM, van Beurden M, Roeters van Lennep JE, van Doorn HC, de Hullu JA, Mom C, van Dorst EBL, Mourits MJE, Slangen BFM, Gaarenstroom KN, Zillikens MC, Leiner T, van der Kolk L, Collee M, Wevers M, Ausems MGEM, van Engelen K, Berger LP, van Asperen CJ, Gomez-Garcia EB, van de Beek I, Rookus MA, Hauptmann M, Bleiker EM, Schagen SB, Aaronson NK, Maas AHEM, van Leeuwen FE. Long-Term Morbidity and Health After Early Menopause Due to Oophorectomy in Women at Increased Risk of Ovarian Cancer: Protocol for a Nationwide Cross-Sectional Study With Prospective Follow-Up (HARMOny Study). JMIR Res Protoc. 2021 Jan 22;10(1):e24414. doi: 10.2196/24414. PMID 33480862